CLINICAL TRIAL: NCT05025098
Title: Precision Therapy Versus Standard Therapy in Acute Myeloid Leukaemia and Myelodysplastic Syndrome in Elderly
Brief Title: Precision Therapy Versus Standard Therapy in AML and MDS in Elderly
Acronym: PALM
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Anders Erik Astrup Dahm, Principal investigator, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PALM
Record Dates: First submitted 2021-05-27; First posted 2021-08-27 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: AML, Adult; MDS
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Standard of Care; Azacitidine; venetoclax

STUDY DESIGN:
Intervention Model Description: randomized open label clinical study phase II
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Standard therapy (Active Comparator): This study is a randomization between treatment principles, not treatments, i.e., standard therapy vs precision therapy (tumor board determined).
  Standard treatment for AML patients is Azacitidine + Venetoclax.*
  *Only if venetoclax is available to the study at the time-point of study start. If venetoclax is not available AML patients will receive Azacitidine alone similar to MDS patients.
  Standard treatment for MDS is Azacitidine.
  Interventions: Drug: Standard therapy
- Precision therapy (Experimental): This study is a randomization between treatment principles, not treatments, i.e., standard therapy vs precision therapy (tumor board determined). The precision therapy arm will receive standard therapy + tumor board decided precision therapy. The tumor board decided precision therapy can in principle be any therapy with marketing authorization in Norway.
  Interventions: Drug: Standard therapy; Drug: Precision therapy

INTERVENTIONS:
Drug: Standard therapy — For AML patients: Venetoclax will be administered orally once daily Days 1 through 28, of a 28-day cycle, with a designated dose of 400 mg daily after ramp up in Cycle 1. During Cycle 1 Days 1 - 3, the dose of Venetoclax will ramp up from 100 mg on Day 1, 200 mg on Day 2, and 400 mg on Day 3. Azacitidine (100 mg/m2) is given once daily following administration of venetoclax for 5 days of every cycle, starting on Day 1 of each cycle.
  For MDS patients: Azacitidine (100 mg/m2) is given once daily for 5 days of every 28 day cycle, starting on day 1 of each cycle.
  Other Names: Azacitidine + venetoclax for AML patients. Azacitidine for MDS patients.
Drug: Precision therapy — Precision therapy for both AML and MDS patients is standard therapy + tumor board determined precision therapy. The tumor board determined precision therapy can be all available drugs with a marketing authorization in Norway.
  Other Names: Standard therapy + tumor board decided precision therapy drug.
  Arms: Precision therapy

SUMMARY:
This is a randomized clinical trial that randomizes between treatment principles. The study will investigate if precision therapy determined by a tumour board is better than standard treatment for acute myeloid leukaemia (AML) and myelodysplastic syndrome (MDS) in elderly. The tumour board will decide the precision therapy based on identified genetic changes that can guide customized therapy. There are currently 40-50 targeted therapies approved for various cancers in Norway. The precision therapy will be given in addition to the standard treatment.

The primary study objective will be to evaluate the cost-effectiveness of a precision therapy strategy compared with standard treatment. Other objectives will mesaure efficacy and satety of the treatment, and impact on life quality of the patients.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) and high-risk myelodysplastic syndrome (MDS) in the elderly are not curable since elderly patients usually do not tolerate intensive chemotherapy and allogeneic stemcell transplantation. Next generation sequencing (NGS) of DNA can find changes in tumor DNA that can be targeted by new drugs, so called "precision therapy". Precision therapy drugs are usually less toxic than standard treatment, and thus may be particularly well suited for elderly. Precision therapy is principally different from today's standard therapy since it will be individualized based on NGS from the tumor, while in standard therapy all patients receive the same treatment. It is unknown how a precision therapy strategy will perform compared with standard therapy in AML and high-risk MDS in the elderly. A Clinical Tumour Board will decide on the precision therapy.

Study design:

This is a prospective, open label, single centre, randomized phase II clinical trial. The study randomizes between standard treatment and precision therapy in unfit elderly patients with AML and high-risk MDS. Importantly, this study design is not a randomization between treatments as in a traditional clinical trial, but a randomization between treatment principles. This means that patients in the standard treatment arm will receive the same treatment, while patients in the precision arm will receive different treatments based on the profiling of the tumor cells. Since most of the precision therapies will be experimental, the study is designed so that the patients in both arms receive a period of standard treatment before randomization. This is to reduce the risk of patients not receiving effective treatment, so that the precision therapy can be tested safely. The standard treatment for AML and high-risk MDS in elderly may change during the study, therefore "standard treatment" is defined as the recommended treatment in Norway at any time point. This means that MDS patients and AML patients may have different standard therapy.

Diagnostic sampling and genomic profiling will be done on the bone marrow of all included patients before start of treatment and compared with germline DNA from buccal swab taken at the bone-marrow. Treatment with hydroxyurea prior to the initial standard treatment is allowed to get leukocytes below 30.

While the patient receive two initial 28 day cycles of standard treatment, NGS of the bone marrow samples are done and assessed in the diagnostic pipeline, followed by bioinformatics analysis. The information is then interpreted by a Clinical Tumour Board consisting of pathologists, haematologists, oncologists, molecular biologists and bioinformatician, the treating hematologist and study nurse. The Clinical Tumour Board makes the decision on targeted treatment.

After initial standard therapy bone marrow samples will be evaluated for response to treatment. Patients with progressive disease as defined by the European Leukemia Net will go out of the study and receive treatment according to investigators choice. Notably, the results from the Clinical Tumour Board will be available for these patients to provide best possible treatment.

Patients without disease progression are randomized in a stratified manner 2:1 after the initial treatment with standard therapy to either precision therapy advised by the Clinical Tumour Board or continuous standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a diagnosis of AML and related precursor neoplasms according to WHO 2016 classification (excluding acute promyelocytic leukemia) including secondary AML (after an antecedent hematological disease and therapy-related AML (not if they have received antileukemic/mds treatment)), or
* acute leukemias of ambiguous lineage according to WHO 2016 or a diagnosis of myelodysplastic syndrome (MDS) with IPSS-R > 4.5.1
* Patients 60 years and older.
* Patients must NOT be eligible for intensive chemotherapy or allogeneic stem cell therapy (See Chapter 23.3)
* WBC ≤ 25 x109/L (prior hydroxyurea allowed for a maximum of 14 days, stopped before start of treatment)
* Adequate renal and hepatic functions unless clearly disease related as indicated by the following laboratory values:
* WHO performance status 0, 1 or 2 for subjects ≥ 75 years of age OR 0 to 3 for subjects ≥ 60 to 74 years of age.
* Life-expectancy above 3 months
* Signed Informed Conscent
* Male Subjects Only: Male subjects who are sexually active, must agree, from Study Day 1 through at least 90 days after the last dose of study drug, to practice contraception with condom. Male subjects must agree to refrain from sperm donation from initial study drug administration until at least 90 days after the last dose of study drug.

Exclusion Criteria:

* Acute promyelocytic leukemia.
* AML with favourable cytogenetic or genetic changes in patients who are fit for intensive chemotherapy. Favourable genetics are: t(8;21)(q22;q22.1); RUNX1-RUNX1T1; inv(16)(p13.1q22) or t(16;16)(p13.1;q22); CBFB-MYH11; mutated NPM1 without FLT3-ITD or with FLT3-ITDlow†; Biallelic mutated CEBPA
* Patients previously treated for AML or MDS (any antileukemic therapy or MDS treatment including investigational agents).
* Patients where it is not possible to get bone-marrow for NGS, i.e., "dry tap".
* Diagnosis of any previous or concomitant malignancy is an exclusion criterion: except when the patient completed successfully treatment (chemotherapy and/or surgery and/or radiotherapy) with curative intent for this malignancy at least 6 months prior to randomization.
* Blast crisis of chronic myeloid leukemia.
* Concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, infection, hypertension, pulmonary disease etc.)
* Cardiac dysfunction as defined by:

  * Unstable angina or
  * New York Heart Association Class ≥ 2. Class 2 is defined as cardiac disease in which patients are comfortable at rest but ordinary physical activity results in fatigue,palpitations, dyspnea, or angina pain or
  * Unstable cardiac arrhythmias
* Patients with a history of non-compliance to medical regimens or who are considered unreliable with respect to compliance with the study protocol and follow-up schedule.
* Patients who have senile dementia, mental impairment or any other psychiatric disorder that prohibits the patient from understanding and giving informed consent.
* Patients who do not understand the Written Informed Consent (e.g., language problems)
* Current concomitant chemotherapy, radiation therapy, or immunotherapy; other than hydroxyurea.
* Subject is known to be positive for HIV (HIV testing is not required).
* Subject is known to be positive for hepatitis B or C infection with the exception of those with an undetectable viral load within 3 months. (Hepatitis B or C testing is not required).
* AML subjects that has received strong and/or moderate CYP3A inducers within 7 days prior to the initiation of venetoclax treatment.
* Subject has a malabsorption syndrome or other condition that precludes enteral route of administration. Additional exclusion criteria at the time of randomization
* WHO performance status > 2 for subjects ≥ 75 years of age OR > 3 for subjects ≥ 60 to 74 years of age.
* Progressive disease according to ELN criteria (see chapter 12 Response evaluation)
* Initial treatment has made the patient eligible for allogeneic stemcell transplantation
* In addition, it will be specific exclusion criteria for the patients receiving targeted therapies related to the Summary of Product Characteristics (SPC) of each drug.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2021-06-22 (Actual); Primary Completion 2026-06-10 (Estimated); Study Completion 2027-06-10 (Estimated)

PRIMARY OUTCOMES:
cost-effectiveness of a precision therapy | 4-5 years
  To evaluate the cost-effectiveness of a precision therapy strategy compared with standard treatment. The total cost of the treatment will be calculated and divided on health related quality of life (HRQoL)

SECONDARY OUTCOMES:
Event free survival | 4-5 years
  Median event free survival, i.e., the number of days to death or progression of the disease (whichever comes first)with AML or MDS
Overall survival | 4-5 years
  Median overall survival
Adverse events | 4-5 years
  The number of adverse events.
Toxicity | 4-5 years
  The number of adverse events with CTCAE grade 3 or more
Transfusion independence | 4-5 years
  The number of erythrocyte- or thrombocyte-transfusionsCR: Bone marrow blasts < 5%; absence of blasts with Auer rods; absence of extramedullary disease; absolute neutrophil count >1.0 x 109/L; platelet count >100 x 109/L
  CR with incomplete recovery (CRi):
  All CR criteria except for residual neutropenia (<1.0 x 109/L) or thrombocytopenia (<100 x 109/L) PR:All hematologic criteria of CR; decrease of bone marrow blast percentage to 5% to 25%; and decrease of pretreatment bone marrow blast percentage by at least 50%
Budget impact | 4-5 years
  Budget impact of providing targeted treatment to all eligible patients.
Overall response rate | 4-5 years
  For AML overall response rate is defined as Complete remission (CR), CR with incomplete recovery (CRi), Morphologic leukemia-free state, or Partial remission. For MDS overall response rate is defined as Complete remission, Marrow Complete Response, or Partial remission.
Quality of life | 4-5 years
  Difference in quality of life using EQ-5D questionnaire between treatment arms
Total costs | 4-5 years
  Total costs of precision therapy.
Progression | 4-5 years
  Median number of days to progression of MDS to AML.
Sequencing quality | 4-5 years
  The fraction of sequencing results with quality good enough to make a decision.
Dry tap | 4-5 years
  The fraction of patients who were excluded because of dry-tap.
Person staff time | 4-5 years
  Person-time used to sequence
Person-time used to find possible precision therapy | 4-5 years
  Person time on tumour board and preparations
Patients with actionable targets | 4-5 years
  The fraction of patients with actionable targets.
MDS progression to AML | 4-5 years
  The median time to AML progression for patients with MDS

CONTACTS AND LOCATIONS:
Overall Officials: Anders Erik Astrup Dahm, MD, PHD, Principal Investigator — Akershus universitetssykehus
Locations (1):
- Akershus Universitetssykehus, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pfeilstocker M, Tuechler H, Sanz G, Schanz J, Garcia-Manero G, Sole F, Bennett JM, Bowen D, Fenaux P, Dreyfus F, Kantarjian H, Kuendgen A, Malcovati L, Cazzola M, Cermak J, Fonatsch C, Le Beau MM, Slovak ML, Levis A, Luebbert M, Maciejewski J, Machherndl-Spandl S, Magalhaes SM, Miyazaki Y, Sekeres MA, Sperr WR, Stauder R, Tauro S, Valent P, Vallespi T, van de Loosdrecht AA, Germing U, Haase D, Greenberg PL. Time-dependent changes in mortality and transformation risk in MDS. Blood. 2016 Aug 18;128(7):902-10. doi: 10.1182/blood-2016-02-700054. Epub 2016 Jun 22. PMID 27335276
- [Background] Lowenberg B, Ossenkoppele GJ, van Putten W, Schouten HC, Graux C, Ferrant A, Sonneveld P, Maertens J, Jongen-Lavrencic M, von Lilienfeld-Toal M, Biemond BJ, Vellenga E, van Marwijk Kooy M, Verdonck LF, Beck J, Dohner H, Gratwohl A, Pabst T, Verhoef G; Dutch-Belgian Cooperative Trial Group for Hemato-Oncology (HOVON); German AML Study Group (AMLSG); Swiss Group for Clinical Cancer Research (SAKK) Collaborative Group. High-dose daunorubicin in older patients with acute myeloid leukemia. N Engl J Med. 2009 Sep 24;361(13):1235-48. doi: 10.1056/NEJMoa0901409. PMID 19776405
- [Background] Burnett A, Wetzler M, Lowenberg B. Therapeutic advances in acute myeloid leukemia. J Clin Oncol. 2011 Feb 10;29(5):487-94. doi: 10.1200/JCO.2010.30.1820. Epub 2011 Jan 10. PMID 21220605
- [Background] Klepin HD, Rao AV, Pardee TS. Acute myeloid leukemia and myelodysplastic syndromes in older adults. J Clin Oncol. 2014 Aug 20;32(24):2541-52. doi: 10.1200/JCO.2014.55.1564. PMID 25071138
- [Background] Klepin HD. Geriatric perspective: how to assess fitness for chemotherapy in acute myeloid leukemia. Hematology Am Soc Hematol Educ Program. 2014 Dec 5;2014(1):8-13. doi: 10.1182/asheducation-2014.1.8. Epub 2014 Nov 18. PMID 25696829
- [Background] Dombret H, Seymour JF, Butrym A, Wierzbowska A, Selleslag D, Jang JH, Kumar R, Cavenagh J, Schuh AC, Candoni A, Recher C, Sandhu I, Bernal del Castillo T, Al-Ali HK, Martinelli G, Falantes J, Noppeney R, Stone RM, Minden MD, McIntyre H, Songer S, Lucy LM, Beach CL, Dohner H. International phase 3 study of azacitidine vs conventional care regimens in older patients with newly diagnosed AML with >30% blasts. Blood. 2015 Jul 16;126(3):291-9. doi: 10.1182/blood-2015-01-621664. Epub 2015 May 18. PMID 25987659
- [Background] Ma X. Epidemiology of myelodysplastic syndromes. Am J Med. 2012 Jul;125(7 Suppl):S2-5. doi: 10.1016/j.amjmed.2012.04.014. PMID 22735748
- [Background] Platzbecker U. Treatment of MDS. Blood. 2019 Mar 7;133(10):1096-1107. doi: 10.1182/blood-2018-10-844696. Epub 2019 Jan 22. PMID 30670446
- [Background] Fenaux P, Mufti GJ, Hellstrom-Lindberg E, Santini V, Finelli C, Giagounidis A, Schoch R, Gattermann N, Sanz G, List A, Gore SD, Seymour JF, Bennett JM, Byrd J, Backstrom J, Zimmerman L, McKenzie D, Beach C, Silverman LR; International Vidaza High-Risk MDS Survival Study Group. Efficacy of azacitidine compared with that of conventional care regimens in the treatment of higher-risk myelodysplastic syndromes: a randomised, open-label, phase III study. Lancet Oncol. 2009 Mar;10(3):223-32. doi: 10.1016/S1470-2045(09)70003-8. Epub 2009 Feb 21. PMID 19230772
- [Background] Prasad V, Gale RP. Precision medicine in acute myeloid leukemia: Hope, hype or both? Leuk Res. 2016 Sep;48:73-7. doi: 10.1016/j.leukres.2016.07.011. Epub 2016 Jul 22. PMID 27497757
- [Background] Hong DS, Bauer TM, Lee JJ, Dowlati A, Brose MS, Farago AF, Taylor M, Shaw AT, Montez S, Meric-Bernstam F, Smith S, Tuch BB, Ebata K, Cruickshank S, Cox MC, Burris HA 3rd, Doebele RC. Larotrectinib in adult patients with solid tumours: a multi-centre, open-label, phase I dose-escalation study. Ann Oncol. 2019 Feb 1;30(2):325-331. doi: 10.1093/annonc/mdy539. PMID 30624546
- [Background] Iyer G, Hanrahan AJ, Milowsky MI, Al-Ahmadie H, Scott SN, Janakiraman M, Pirun M, Sander C, Socci ND, Ostrovnaya I, Viale A, Heguy A, Peng L, Chan TA, Bochner B, Bajorin DF, Berger MF, Taylor BS, Solit DB. Genome sequencing identifies a basis for everolimus sensitivity. Science. 2012 Oct 12;338(6104):221. doi: 10.1126/science.1226344. Epub 2012 Aug 23. PMID 22923433
- [Background] Ree AH, Nygaard V, Russnes HG, Heinrich D, Nygaard V, Johansen C, Bergheim IR, Hovig E, Beiske K, Negard A, Borresen-Dale AL, Flatmark K, Maelandsmo GM. Responsiveness to PD-1 Blockade in End-Stage Colon Cancer with Gene Locus 9p24.1 Copy-Number Gain. Cancer Immunol Res. 2019 May;7(5):701-706. doi: 10.1158/2326-6066.CIR-18-0777. Epub 2019 Feb 25. PMID 30804006
- [Background] Von Hoff DD, Stephenson JJ Jr, Rosen P, Loesch DM, Borad MJ, Anthony S, Jameson G, Brown S, Cantafio N, Richards DA, Fitch TR, Wasserman E, Fernandez C, Green S, Sutherland W, Bittner M, Alarcon A, Mallery D, Penny R. Pilot study using molecular profiling of patients' tumors to find potential targets and select treatments for their refractory cancers. J Clin Oncol. 2010 Nov 20;28(33):4877-83. doi: 10.1200/JCO.2009.26.5983. Epub 2010 Oct 4. PMID 20921468
- [Background] Tyner JW, Tognon CE, Bottomly D, Wilmot B, Kurtz SE, Savage SL, Long N, Schultz AR, Traer E, Abel M, Agarwal A, Blucher A, Borate U, Bryant J, Burke R, Carlos A, Carpenter R, Carroll J, Chang BH, Coblentz C, d'Almeida A, Cook R, Danilov A, Dao KT, Degnin M, Devine D, Dibb J, Edwards DK 5th, Eide CA, English I, Glover J, Henson R, Ho H, Jemal A, Johnson K, Johnson R, Junio B, Kaempf A, Leonard J, Lin C, Liu SQ, Lo P, Loriaux MM, Luty S, Macey T, MacManiman J, Martinez J, Mori M, Nelson D, Nichols C, Peters J, Ramsdill J, Rofelty A, Schuff R, Searles R, Segerdell E, Smith RL, Spurgeon SE, Sweeney T, Thapa A, Visser C, Wagner J, Watanabe-Smith K, Werth K, Wolf J, White L, Yates A, Zhang H, Cogle CR, Collins RH, Connolly DC, Deininger MW, Drusbosky L, Hourigan CS, Jordan CT, Kropf P, Lin TL, Martinez ME, Medeiros BC, Pallapati RR, Pollyea DA, Swords RT, Watts JM, Weir SJ, Wiest DL, Winters RM, McWeeney SK, Druker BJ. Functional genomic landscape of acute myeloid leukaemia. Nature. 2018 Oct;562(7728):526-531. doi: 10.1038/s41586-018-0623-z. Epub 2018 Oct 17. PMID 30333627
- [Background] Haferlach T, Nagata Y, Grossmann V, Okuno Y, Bacher U, Nagae G, Schnittger S, Sanada M, Kon A, Alpermann T, Yoshida K, Roller A, Nadarajah N, Shiraishi Y, Shiozawa Y, Chiba K, Tanaka H, Koeffler HP, Klein HU, Dugas M, Aburatani H, Kohlmann A, Miyano S, Haferlach C, Kern W, Ogawa S. Landscape of genetic lesions in 944 patients with myelodysplastic syndromes. Leukemia. 2014 Feb;28(2):241-7. doi: 10.1038/leu.2013.336. Epub 2013 Nov 13. PMID 24220272
- [Background] Stone RM, Mandrekar SJ, Sanford BL, Laumann K, Geyer S, Bloomfield CD, Thiede C, Prior TW, Dohner K, Marcucci G, Lo-Coco F, Klisovic RB, Wei A, Sierra J, Sanz MA, Brandwein JM, de Witte T, Niederwieser D, Appelbaum FR, Medeiros BC, Tallman MS, Krauter J, Schlenk RF, Ganser A, Serve H, Ehninger G, Amadori S, Larson RA, Dohner H. Midostaurin plus Chemotherapy for Acute Myeloid Leukemia with a FLT3 Mutation. N Engl J Med. 2017 Aug 3;377(5):454-464. doi: 10.1056/NEJMoa1614359. Epub 2017 Jun 23. PMID 28644114
- [Background] Cortes JE, Tallman MS, Schiller GJ, Trone D, Gammon G, Goldberg SL, Perl AE, Marie JP, Martinelli G, Kantarjian HM, Levis MJ. Phase 2b study of 2 dosing regimens of quizartinib monotherapy in FLT3-ITD-mutated, relapsed or refractory AML. Blood. 2018 Aug 9;132(6):598-607. doi: 10.1182/blood-2018-01-821629. Epub 2018 Jun 6. PMID 29875101
- [Background] Stein EM, DiNardo CD, Fathi AT, Pollyea DA, Stone RM, Altman JK, Roboz GJ, Patel MR, Collins R, Flinn IW, Sekeres MA, Stein AS, Kantarjian HM, Levine RL, Vyas P, MacBeth KJ, Tosolini A, VanOostendorp J, Xu Q, Gupta I, Lila T, Risueno A, Yen KE, Wu B, Attar EC, Tallman MS, de Botton S. Molecular remission and response patterns in patients with mutant-IDH2 acute myeloid leukemia treated with enasidenib. Blood. 2019 Feb 14;133(7):676-687. doi: 10.1182/blood-2018-08-869008. Epub 2018 Dec 3. PMID 30510081
- [Background] Cerrano M, Itzykson R. New Treatment Options for Acute Myeloid Leukemia in 2019. Curr Oncol Rep. 2019 Feb 4;21(2):16. doi: 10.1007/s11912-019-0764-8. PMID 30715623
- [Background] Welch JS, Petti AA, Miller CA, Fronick CC, O'Laughlin M, Fulton RS, Wilson RK, Baty JD, Duncavage EJ, Tandon B, Lee YS, Wartman LD, Uy GL, Ghobadi A, Tomasson MH, Pusic I, Romee R, Fehniger TA, Stockerl-Goldstein KE, Vij R, Oh ST, Abboud CN, Cashen AF, Schroeder MA, Jacoby MA, Heath SE, Luber K, Janke MR, Hantel A, Khan N, Sukhanova MJ, Knoebel RW, Stock W, Graubert TA, Walter MJ, Westervelt P, Link DC, DiPersio JF, Ley TJ. TP53 and Decitabine in Acute Myeloid Leukemia and Myelodysplastic Syndromes. N Engl J Med. 2016 Nov 24;375(21):2023-2036. doi: 10.1056/NEJMoa1605949. PMID 27959731
- [Background] Lambert J, Pautas C, Terre C, Raffoux E, Turlure P, Caillot D, Legrand O, Thomas X, Gardin C, Gogat-Marchant K, Rubin SD, Benner RJ, Bousset P, Preudhomme C, Chevret S, Dombret H, Castaigne S. Gemtuzumab ozogamicin for de novo acute myeloid leukemia: final efficacy and safety updates from the open-label, phase III ALFA-0701 trial. Haematologica. 2019 Jan;104(1):113-119. doi: 10.3324/haematol.2018.188888. Epub 2018 Aug 3. PMID 30076173
- [Background] Cortizas EM, Zahn A, Safavi S, Reed JA, Vega F, Di Noia JM, Verdun RE. UNG protects B cells from AID-induced telomere loss. J Exp Med. 2016 Oct 17;213(11):2459-2472. doi: 10.1084/jem.20160635. Epub 2016 Oct 3. PMID 27697833
- [Background] Fountzilas E, Tsimberidou AM. Overview of precision oncology trials: challenges and opportunities. Expert Rev Clin Pharmacol. 2018 Aug;11(8):797-804. doi: 10.1080/17512433.2018.1504677. Epub 2018 Aug 10. PMID 30044653
- [Background] Le Tourneau C, Delord JP, Goncalves A, Gavoille C, Dubot C, Isambert N, Campone M, Tredan O, Massiani MA, Mauborgne C, Armanet S, Servant N, Bieche I, Bernard V, Gentien D, Jezequel P, Attignon V, Boyault S, Vincent-Salomon A, Servois V, Sablin MP, Kamal M, Paoletti X; SHIVA investigators. Molecularly targeted therapy based on tumour molecular profiling versus conventional therapy for advanced cancer (SHIVA): a multicentre, open-label, proof-of-concept, randomised, controlled phase 2 trial. Lancet Oncol. 2015 Oct;16(13):1324-34. doi: 10.1016/S1470-2045(15)00188-6. Epub 2015 Sep 3. PMID 26342236
- [Background] DiNardo CD, Pratz K, Pullarkat V, Jonas BA, Arellano M, Becker PS, Frankfurt O, Konopleva M, Wei AH, Kantarjian HM, Xu T, Hong WJ, Chyla B, Potluri J, Pollyea DA, Letai A. Venetoclax combined with decitabine or azacitidine in treatment-naive, elderly patients with acute myeloid leukemia. Blood. 2019 Jan 3;133(1):7-17. doi: 10.1182/blood-2018-08-868752. Epub 2018 Oct 25. PMID 30361262
- [Background] Wei AH, Montesinos P, Ivanov V, DiNardo CD, Novak J, Laribi K, Kim I, Stevens DA, Fiedler W, Pagoni M, Samoilova O, Hu Y, Anagnostopoulos A, Bergeron J, Hou JZ, Murthy V, Yamauchi T, McDonald A, Chyla B, Gopalakrishnan S, Jiang Q, Mendes W, Hayslip J, Panayiotidis P. Venetoclax plus LDAC for newly diagnosed AML ineligible for intensive chemotherapy: a phase 3 randomized placebo-controlled trial. Blood. 2020 Jun 11;135(24):2137-2145. doi: 10.1182/blood.2020004856. PMID 32219442
- [Background] DiNardo CD, Jonas BA, Pullarkat V, Thirman MJ, Garcia JS, Wei AH, Konopleva M, Dohner H, Letai A, Fenaux P, Koller E, Havelange V, Leber B, Esteve J, Wang J, Pejsa V, Hajek R, Porkka K, Illes A, Lavie D, Lemoli RM, Yamamoto K, Yoon SS, Jang JH, Yeh SP, Turgut M, Hong WJ, Zhou Y, Potluri J, Pratz KW. Azacitidine and Venetoclax in Previously Untreated Acute Myeloid Leukemia. N Engl J Med. 2020 Aug 13;383(7):617-629. doi: 10.1056/NEJMoa2012971. PMID 32786187
- [Background] Burd A. Initial Report of the Beat AML Umbrella Study for Previously Untreated AML: Evidence of Feasibility and Early Success in Molecularly Driven Phase 1 and 2 studies. Annual meeting of the American Society of Hematology. San Diego; 2018
- [Background] Dohner H, Estey E, Grimwade D, Amadori S, Appelbaum FR, Buchner T, Dombret H, Ebert BL, Fenaux P, Larson RA, Levine RL, Lo-Coco F, Naoe T, Niederwieser D, Ossenkoppele GJ, Sanz M, Sierra J, Tallman MS, Tien HF, Wei AH, Lowenberg B, Bloomfield CD. Diagnosis and management of AML in adults: 2017 ELN recommendations from an international expert panel. Blood. 2017 Jan 26;129(4):424-447. doi: 10.1182/blood-2016-08-733196. Epub 2016 Nov 28. PMID 27895058
- [Background] Cheson BD, Greenberg PL, Bennett JM, Lowenberg B, Wijermans PW, Nimer SD, Pinto A, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Gore SD, Schiffer CA, Kantarjian H. Clinical application and proposal for modification of the International Working Group (IWG) response criteria in myelodysplasia. Blood. 2006 Jul 15;108(2):419-25. doi: 10.1182/blood-2005-10-4149. Epub 2006 Apr 11. PMID 16609072
- [Background] Arber DA, Orazi A, Hasserjian R, et al. The 2016 revision to the World Health Organization classification of myeloid neoplasms and acute leukemia. Blood. 2016;127(20):2391-2405. Blood. 2016 Jul 21;128(3):462-463. doi: 10.1182/blood-2016-06-721662. No abstract available. PMID 31659364
- [Background] Li MM, Datto M, Duncavage EJ, Kulkarni S, Lindeman NI, Roy S, Tsimberidou AM, Vnencak-Jones CL, Wolff DJ, Younes A, Nikiforova MN. Standards and Guidelines for the Interpretation and Reporting of Sequence Variants in Cancer: A Joint Consensus Recommendation of the Association for Molecular Pathology, American Society of Clinical Oncology, and College of American Pathologists. J Mol Diagn. 2017 Jan;19(1):4-23. doi: 10.1016/j.jmoldx.2016.10.002. PMID 27993330